CLINICAL TRIAL: NCT06687460
Title: Brief Electrical Stimulation for Promoting Peripheral Nerve Regeneration After Primary Neurorrhaphy of Upper Extremities
Brief Title: Distal Nerve Electrical Stimulation for Neuromuscular Reinnervation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-112-085
Record Dates: First submitted 2024-11-05; First posted 2024-11-13 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-07

CONDITIONS: Electrical Stimulation; Peripheral Nerve Regeneration
Keywords: electrical stimulation; peripheral nerve regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nerve electrical stimulation (Experimental): During the process of nerve microsurgical reconstruction, a 30-minute electric stimulation is applied to the distal end of the damaged nerve.
  Interventions: Other: Brief electrical stimulation
- nerve microsurgical reconstruction (Placebo Comparator): no nerve electrical stimulation
  Interventions: Other: no nerve electrical stimulation

INTERVENTIONS:
Other: Brief electrical stimulation — During the nerve micro-reconstruction surgery, electrical stimulation is given to the distal end of the damaged nerve for 30 minutes.
  Arms: nerve electrical stimulation
Other: no nerve electrical stimulation — only nerve microsurgical reconstruction, no nerve electrical stimulation
  Arms: nerve microsurgical reconstruction

SUMMARY:
During the process of nerve microsurgical reconstruction, 30 minutes of electrical stimulation is applied to the distal end of the damaged nerve to assess its potential benefits for nerve regeneration, functional recovery, slowing down the degeneration at the neuromuscular junction, and preventing muscle atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Acute peripheral nerve rupture between the elbow and wrist
* Acute rupture of the median or ulnar nerve
* Patients who have signed a valid written consent for surgery and trials

Exclusion Criteria:

* History of injury or other causes leading to muscle and joint dysfunction in the affected area
* Patients with radial nerve damage
* Diabetes
* History of arrhythmia
* Stroke
* Multiple sclerosis
* Hereditary peripheral neuropathy
* Amyotrophic lateral sclerosis (ALS)
* Patients with a pacemaker
* Presence of local infection at the wound site
* Pregnant or breastfeeding women
* Patients deemed unsuitable for enrollment by a physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
NCV/EMG(CMAP,latency) | The third month after surgery.
  The electromyography (EMG) is a diagnostic method used to assess muscle and nerve function, primarily to detect muscle activity and nerve conduction velocity, in order to monitor the recovery of neuromuscular function after surgery. During the EMG examination, the examiner uses electrodes attached to the palm to measure and record the electrophysiological signals of the muscles for further analysis. Through this method, doctors can evaluate the electrophysiological activity of the muscles to assess the reinnervation of distal muscles by the damaged nerves.

SECONDARY OUTCOMES:
DASH questionnaire | The first, third, and sixth months after surgery.
  The DASH questionnaire (Disabilities of the Arm, Shoulder, and Hand) is a tool used to assess a patient's upper extremity function and symptoms. It helps in evaluating the impact of musculoskeletal disorders on daily activities and quality of life.
Muscle power | The third and sixth months after surgery.
  Muscle power refers to the ability of a muscle or group of muscles to exert force quickly. It is a combination of strength and speed, and is often measured in activities that require explosive movements, such as sprinting, jumping, or lifting weights. Muscle power is important for athletic performance and functional movement in daily activities.
Purdue Pegboard test | The third and sixth months after surgery.
  The Purdue Pegboard test is a standardized assessment used to measure manual dexterity and fine motor skills. It involves placing pegs into holes on a board as quickly and accurately as possible, using one hand at a time and then both hands. The test is commonly used in occupational therapy, rehabilitation, and research to evaluate hand function and coordination.
MMDT | The third and sixth months after surgery
  Assessment of hand dexterity and posture tolerance
NCV/EMG(CMAP,latency) | The sixth month after surgery.
  Electromyography (EMG) is a diagnostic method used to assess muscle and nerve function, primarily for detecting muscle activity and nerve conduction velocity to monitor the recovery of neuromuscular function post-surgery. During an EMG examination, the examiner attaches electrodes to the palm to measure and record the electrophysiological signals of the muscles for further analysis. This allows physicians to evaluate the electrophysiological activity of the muscles and assess the reinnervation of distal muscles by the damaged nerves.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan, Taiwan